CLINICAL TRIAL: NCT07233278
Title: Effects of High-Intensity, Low-Frequency Periodic rTMS Over the Right Dorsolateral Prefrontal Cortex on Cardiac Autonomic Regulation in Women With Recurrent Pregnancy Loss and Anxiety: A Randomized, Sham-Controlled, Proof-of-Concept Trial (NEURO-CARD-rTMS-2)
Brief Title: High-Intensity, Low-Frequency Periodic rTMS Over the Right Dorsolateral Prefrontal Cortex on Cardiac Autonomic Regulation in Women With Recurrent Pregnancy Loss and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenyang Medical College (Other)
Collaborators: Central Hospital Affiliated to Shenyang Medical Collage (Other); The Second Hospital of Shenyang Medical College (Other)
Responsible Party: Principal Investigator, Lin Tao, Assoc.Prof., Shenyang Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-038-02
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Pregnancy Loss(RPL); Anxiety
Keywords: Recurrent pregnancy loss; Anxiety; Dorsolateral Prefrontal Cortex; Cardiac Autonomic Regulation; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study will use a parallel assignment interventional model. Participants will be randomly assigned in a 1:1 ratio to either the active rTMS group or the sham rTMS group. Each participant will receive a single-session intervention under their assigned condition. The intervention will be delivered in a controlled laboratory setting, and both groups will undergo identical procedures except for the presence or absence of effective magnetic stimulation. This design allows for between-group comparison of physiological responses and safety outcomes attributable to the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will remain blinded to group allocation throughout the study. Only the rTMS operators will be aware of the intervention assignment, as they are responsible for administering either active or sham stimulation. Sham stimulation will be delivered using a 45°-angled coil to replicate the scalp sensations of active rTMS while minimizing cortical effects. All data labeling, processing, and statistical analysis will be conducted under blinded conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real rTMS group (Active Comparator): Participants in this arm will receive active repetitive transcranial magnetic stimulation (rTMS) delivered to the right dorsolateral prefrontal cortex (DLPFC). The stimulation protocol consists of 20 consecutive cycles of low-frequency (1 Hz) rTMS at 120% of the resting motor threshold (RMT), with each cycle comprising 40 seconds of stimulation followed by 20 seconds of rest. The total stimulation duration is approximately 20 minutes. Real stimulation is applied with the figure-eight coil positioned tangentially to the scalp.
  Interventions: Device: Rhythmic repetitive transcranial magnetic stimulation (rTMS) at 120% RMT, 1 Hz, 60-s cycles
- sham rTMS group (Sham Comparator): Participants in this arm will receive sham repetitive transcranial magnetic stimulation (rTMS) over the right dorsolateral prefrontal cortex (DLPFC). The stimulation protocol mimics the active condition in timing and coil placement but involves tilting the coil at a 45-degree angle to the scalp, significantly attenuating magnetic field penetration. This approach preserves the auditory and tactile sensations of stimulation without producing cortical effects. The procedure consists of 20 consecutive cycles of sham stimulation, each comprising 40 seconds of simulated stimulation followed by 20 seconds of rest, lasting approximately 20 minutes in total.
  Interventions: Device: Rhythmic repetitive transcranial magnetic stimulation (rTMS) at 120% RMT, 1 Hz, 60-s cycles

INTERVENTIONS:
Device: Rhythmic repetitive transcranial magnetic stimulation (rTMS) at 120% RMT, 1 Hz, 60-s cycles — Participants in the real rTMS group will receive rhythmic low-frequency repetitive transcranial magnetic stimulation (rTMS) applied over the right dorsolateral prefrontal cortex (DLPFC). The intervention consists of 20 consecutive stimulation cycles, each comprising 40 seconds of 1 Hz stimulation followed by a 20-second inter-cycle interval, totaling 60 seconds per cycle. The stimulation intensity is set at 120% of the individual's resting motor threshold (RMT). A figure-of-eight coil will be positioned tangentially over the scalp at the targeted right DLPFC site. Electrocardiogram (ECG) signals will be recorded synchronously throughout the session for heart rate variability analysis.

SUMMARY:
The goal of this clinical trial is to determine whether high-intensity, low-frequency periodic repetitive transcranial magnetic stimulation (rTMS) applied to the right dorsolateral prefrontal cortex (DLPFC) can modulate cardiac autonomic regulation in women with recurrent pregnancy loss (RPL) and comorbid anxiety. The main questions it aims to answer are:

Does 120% resting motor threshold (RMT) rhythmic low-frequency rTMS reduce heart rate during stimulation time windows compared with sham stimulation?

Does 120% RMT rTMS alter heart-rate-variability (HRV) spectral power at the target frequency (0.0167 Hz) compared with sham stimulation?

Researchers will compare active rTMS with sham rTMS to determine whether the active intervention produces measurable changes in cardiac autonomic activity.

Participants will:

Undergo a single session of rTMS or sham stimulation consisting of 20 consecutive stimulation time windows (each 60 seconds: 40 seconds of 1-Hz stimulation plus 20 seconds of rest) targeting the right DLPFC;

Have continuous electrocardiography (ECG) recordings collected during the entire stimulation session;

Complete clinical and psychiatric assessments before participation.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL), defined as the loss of two or more pregnancies before viability (i.e., 24 weeks by European standards or 28 weeks by Chinese criteria), affects approximately 2-5% of women of reproductive age and represents a significant physical and psychological burden. Beyond its implications for reproductive health, RPL is increasingly recognized as a condition associated with systemic consequences, including heightened anxiety, altered autonomic nervous system function, and increased long-term cardiovascular risk.

Emerging evidence suggests that in women with RPL and comorbid anxiety, chronic psychological stress may lead to dysregulation of the autonomic nervous system, characterized by increased sympathetic tone, reduced vagal activity, elevated resting heart rate, and decreased heart rate variability (HRV). These alterations may create a maladaptive feedback loop that reinforces emotional distress, autonomic imbalance, and reproductive vulnerability.

To address this issue, this randomized, sham-controlled, proof-of-concept clinical trial will investigate whether low-frequency repetitive transcranial magnetic stimulation (rTMS) targeting the right dorsolateral prefrontal cortex (DLPFC)-a region critically involved in emotion regulation and autonomic control-can modulate cardiac autonomic function in women with RPL and anxiety.

The intervention protocol is based on findings from a prior dose-finding study (NEURO-CARD-rTMS-1), which indicated that stimulation at 120% of resting motor threshold (RMT) produced significant reductions in heart rate without compromising tolerability. Building on this, the current trial (NEURO-CARD-rTMS-2) will apply 1-Hz rhythmic rTMS at 120% RMT over the right DLPFC, delivered in 20 consecutive stimulation windows (each 60 seconds long: 40 seconds of stimulation followed by 20 seconds of rest). This stimulation paradigm aligns with the very-low-frequency (VLF) band of HRV (~0.0167 Hz), enabling frequency-specific entrainment analysis.

The primary endpoint will be the difference in baseline-corrected mean heart rate during the stimulation time windows between the active and sham groups. Secondary endpoints include changes in HRV spectral power at 0.0167 Hz and brain-heart coupling (BHC), defined as the correlation between heart rate and spectral power at this frequency. Safety outcomes will be monitored throughout the procedure.

All electrocardiographic (ECG) data will be recorded continuously at 1000 Hz using a wireless Bluetooth system. Participants will undergo standardized psychiatric assessments based on DSM-5 criteria, and key demographic and clinical variables (e.g., BMI, blood pressure, medication use, number and cause of miscarriages) will be collected for covariate analysis.

This trial aims to provide initial mechanistic evidence for the feasibility and physiological efficacy of right DLPFC-targeted neuromodulation in improving autonomic regulation in a high-risk, psychologically sensitive population. If successful, the findings will support the development of non-invasive, brain-based interventions to improve both reproductive and cardiovascular outcomes in women with RPL and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* (i) Female, aged 18-45 years, and right-handed;
* (ii) Diagnosed with recurrent pregnancy loss (RPL), defined as two or more consecutive spontaneous miscarriages occurring before 28 weeks of gestation;
* (iii) Not currently pregnant or in a state of missed miscarriage;
* (iv) Meeting the diagnostic criteria for an anxiety disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).

Exclusion Criteria:

* (i) Contraindications to transcranial magnetic stimulation (TMS), such as metallic implants or a history of epilepsy;
* (ii) Unstable blood pressure (systolic >180 mmHg or <90 mmHg);
* (iii) Coexisting major organic disorders, including hyperthyroidism, atrial fibrillation, valvular heart disease, sinus bradycardia, neurological diseases, cerebrovascular disease, or pulmonary disorders;
* (iv) Significant suicide risk;
* (v) Other psychiatric disorders, including substance use disorders, schizophrenia, delusional disorder, unspecified psychotic disorder, bipolar disorder, or delirium.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the between-group difference in baseline-corrected mean heart rate, averaged across stimulation time windows. | Session 1 (Day 1)
  Heart rate (HR) will be continuously recorded via ECG (1,000 Hz) during a single rTMS session comprising 20 stimulation cycles (each 60 s: 40 s stimulation at 1 Hz, then 20 s rest). For each cycle, a 50-s analysis window will be defined (-10 s to 0 s pre-stimulation baseline; 0 s to +40 s post-stimulation). Baseline-corrected mean HR for each cycle will be computed as the mean HR in the post-stimulation segment (0-40 s) minus the mean HR in the 10-s pre-stimulation baseline (-10-0 s). Per-participant values will then be averaged across the 20 stimulation time windows, and the primary endpoint will compare these averaged baseline-corrected means between the active and sham rTMS groups.

SECONDARY OUTCOMES:
The between-group difference in heart rate variability (HRV) spectral power at the target frequency (0.0167 Hz), averaged across stimulation time windows. | Session 1 (Day 1)
  HRV spectral power at the target frequency will be derived from R-R interval (RRI) series obtained from continuous ECG (1,000 Hz). RRI will be resampled at 1 Hz via cubic-spline interpolation, linearly detrended, and band-pass filtered. Time-frequency analysis will use a derivative-of-Gaussian (DoG) wavelet. For each stimulation cycle (60 s; 40 s stimulation + 20 s rest), a 50-s stimulation time window will be defined (-10 s to +40 s relative to stimulation onset). Frequency-specific entrainment power will be computed as the mean wavelet power within 0.015-0.018 Hz inside this window. Per-participant estimates will then be averaged across the 20 stimulation time windows, and active versus sham groups will be compared.
The strength of the linear correlation (i.e., brain-heart coupling, BHC) between baseline-corrected mean heart rate and spectral power at 0.0167 Hz, averaged across stimulation time windows, in the active rTMS group. | Session 1 (Day 1)
  For each participant in the active rTMS group, the linear correlation (Pearson's r) between these two window-wise measures will be calculated across the 20 stimulation time windows.
The strength of the linear correlation (i.e., BHC) between baseline-corrected mean heart rate and spectral power at 0.0167 Hz, averaged across stimulation time windows, in the sham rTMS group. | Session 1 (Day 1)
  For each participant in the sham rTMS group, the linear correlation (Pearson's r) between these two window-wise measures will be calculated across the 20 stimulation time windows.
Incidence of mild adverse events during rTMS stimulation, including scalp discomfort at the stimulation site, facial muscle twitching, mild headache, and dizziness. | Session 1 (Day 1)
  This outcome will capture the incidence (proportion of participants with ≥1 event) of prespecified mild adverse events during the rTMS session and the immediate 1-hour post-session observation period. Mild events include scalp discomfort at the stimulation site, facial muscle twitching, mild headache, and dizziness. Events will be solicited and recorded in real time by trained operators using a standardized checklist, with participant self-report. Vital signs (blood pressure and resting heart rate) will be reassessed at the end of the session. Events will be classified as mild if transient, self-limited, not requiring medical treatment, and not meeting serious adverse event criteria (e.g., syncope or seizure). Incidence will be summarized by group (active vs sham) for comparison.
Incidence of serious adverse events during rTMS stimulation, including syncope and seizures. | Session 1 (Day 1)
  This outcome will quantify the incidence (proportion of participants with ≥1 event) of serious adverse events (SAEs) occurring during the rTMS session and the subsequent 1-hour observation period. SAEs will be defined per ICH-GCP criteria (events that are fatal, life-threatening, require inpatient hospitalization or prolong an existing hospitalization, result in persistent or significant disability/incapacity, or are otherwise medically important). Events of special interest include syncope and seizures. Trained operators will actively monitor and document SAEs in real time using standardized case-report forms, including onset time, duration, actions taken, outcome, and relatedness to the intervention. Any suspected SAE will trigger protocol-specified safety procedures (immediate termination of stimulation, vital-sign reassessment, medical evaluation, and referral as needed). Incidence will be summarized by group (active vs sham).

CONTACTS AND LOCATIONS:
Overall Officials: Yun-En Liu, MD, Study Chair — Shenyang Medical College; Lin Tao, MM, Principal Investigator — Shenyang Medical College; Fei Meng, MD, Study Director — Central Hospital Affiliated to Shenyang Medical Collage
Locations (1):
- Central Hospital Affiliated to Shenyang Medical Collage, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, study protocol and supporting materials will be made publicly available at the time of formal publication. Data will be hosted on an internationally recognised third-party repository and accessible for non-commercial scientific use.
Supporting Information: Study Protocol
Time Frame: Available at the time of formal publication